CLINICAL TRIAL: NCT03692611
Title: Evaluation of the Efficacy and Mechanisms of a Novel Intervention for Chronic Pain Tailored to People Living With HIV
Acronym: STOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Alabama at Birmingham (Other); National Institute of Mental Health (NIMH) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Jessica Merlin, Visiting Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY19050051; 1R01MH115754-01A1 (NIH)
Record Dates: First submitted 2018-09-07; First posted 2018-10-02 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
Keywords: Chronic pain; HIV; Opioid prescribing; Behavioral clinical trial
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial to discover whether STOMP is an efficacious Pain Self-Management (PSM) intervention, mediated by the hypothesized Social Cognitive Theory (SCT) constructs.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skills to Manage Pain (STOMP) (Experimental): The intervention group will receive treatment as usual plus the STOMP behavioral intervention. The STOMP behavioral intervention consists of 12 intervention sessions (6 group and 6 individual sessions). The sessions will be completed over a period of 12-16 weeks from enrollment. The first intervention session will be a group session for all participants followed by individual and then alternating group and individual sessions for the rest of the intervention. The intervention group will utilize a study manual on pain management in which they will use with each session.
  Interventions: Behavioral: Skills TO Manage Pain (STOMP)
- comparison group (Active Comparator): The comparison group will receive treatment as usual.The comparison group will also be provided with the intervention manual, however, no additional treatment will be provided to participants allocated to the control group. The group will not receive the PSM intervention.
  Interventions: Behavioral: Comparison group

INTERVENTIONS:
Behavioral: Skills TO Manage Pain (STOMP) — 12 week pain self management (PSM) intervention incorporating social cognitive theory constructs.
  Arms: Skills to Manage Pain (STOMP)
Behavioral: Comparison group — Participants in this arm will receive usual care as given by providers but no behavioral PSM intervention.
  Other Names: active comparator
  Arms: comparison group

SUMMARY:
Due to its prevalence and impact on quality of life and overall health, the National Academy of Medicine has called chronic pain a "public health crisis." Therefore, this proposal is relevant to public health because it seeks to improve chronic pain treatment in accordance with the approach recommended by the Department of Health and Human Services National Pain Strategy: to develop and test Pain Self-Management interventions tailored to the needs of vulnerable populations, particularly people living with HIV (PLWH). Chronic pain is an important and understudied comorbidity among PLWH; therefore, this proposal is responsive to the NIH's HIV Research Priorities, which identify comorbidities as a high priority research topic.

DETAILED DESCRIPTION:
Behavioral interventions for chronic pain among people living with HIV (PLWH) are an understudied area, with great potential to improve pain and function. Chronic pain is an important comorbidity that affects between 30% and 85% of PLWH and is associated with greater odds of functional impairment, increased emergency room utilization, suboptimal retention in HIV care, and failure to achieve virologic suppression. What is not known is how to optimally address chronic pain in this population. Opioids are a commonly used treatment for chronic pain, particularly in PLWH. Opioid prescribing for chronic pain often does not result in substantial improvement in outcomes and contributes to the growing epidemic of opioid addiction and overdose. In contrast, behavioral interventions are among the most effective and safest treatments for chronic pain in the general population. Pain Self-Management (PSM) is a Social Cognitive Theory (SCT)-based behavioral approach that involves pain-related skill acquisition and goal setting. PSM interventions have been promoted by the 2016 Department of Health and Human Services National Pain Strategy (DHHS NPS) as an effective, scalable approach to chronic pain management. Especially given the current opioid crisis, the DHHS NPS underscored the urgent need to develop and test PSM interventions tailored to the unique needs of vulnerable populations, particularly PLWH, that can be implemented and disseminated nationwide. Until an effective and scalable PSM intervention for chronic pain in PLWH is developed, reducing the burden of chronic pain safely and effectively in this population will not be possible. The overall objective of this proposal is to evaluate a novel theory-based PSM intervention, "Skills TO Manage Pain" (STOMP), developed for and tailored to PLWH. The investigators will accomplish the overall objective with the following primary specific aim: 1) Evaluate the efficacy of STOMP, a theory-based intervention tailored to improving chronic pain in PLWH. Given the investigators' rigorous intervention development process and promising pilot trial results, the working hypothesis is that STOMP will decrease pain and improve function in PLWH. Investigators also propose the following secondary aims: 2) Conduct exploratory analyses of the impact of STOMP on HIV outcomes associated with chronic pain (i.e. retention in care, virologic suppression), and 3) Investigate proximal outcomes as potential mediators of STOMP's impact on chronic pain. This approach is innovative because it incorporates novel peer co-led group sessions that were created based on the investigators' formative intervention development work, includes patients with comorbidities (e.g., depressive symptoms, addiction history) common among PLWH but typically excluded from chronic pain studies, and investigates the impact of a chronic pain intervention on disease-specific HIV outcomes in addition to pain and function. The proposed research will be significant because if successful, it will pave the way for future dissemination and implementation studies that have the potential to dramatically change chronic pain treatment for PLWH.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in CNICS
2. Age ≥ 18 years
3. English-speaking
4. Chronic pain (Brief Chronic Pain Screening Questionnaire (BCPQ) = at least moderate pain for at least 3 months)
5. Moderately severe and impairing chronic pain (PEG pain questionnaire = average of all three items is 4 or greater)
6. Ability and willingness to attend the group sessions at the date/time specified
7. No plans for major surgery during the study period that would interfere with study procedures.

Exclusion Criteria:

1. Do not speak or understand English
2. Are planning a new pain treatment like surgery
3. Cannot attend the group sessions
4. Had previously participated in the pilot study (STOMP)
5. Unwilling to provide informed consent

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2025-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Merlin, MD PhD MBA, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merlin JS, Westfall AO, Raper JL, Zinski A, Norton WE, Willig JH, Gross R, Ritchie CS, Saag MS, Mugavero MJ. Pain, mood, and substance abuse in HIV: implications for clinic visit utilization, antiretroviral therapy adherence, and virologic failure. J Acquir Immune Defic Syndr. 2012 Oct 1;61(2):164-70. doi: 10.1097/QAI.0b013e3182662215. PMID 22766967
- [Background] Merlin JS, Westfall AO, Johnson MO, Kerns RD, Bair MJ, Kertesz S, Turan JM, Clay OJ, Starrels JL, Kilgore M. Cost-effectiveness of a chronic pain intervention for people living with HIV (PLWH). J Med Econ. 2018 Feb;21(2):122-126. doi: 10.1080/13696998.2017.1377719. Epub 2017 Sep 18. PMID 28880698
- [Background] Merlin JS, Westfall AO, Chamot E, Overton ET, Willig JH, Ritchie C, Saag MS, Mugavero MJ. Pain is independently associated with impaired physical function in HIV-infected patients. Pain Med. 2013 Dec;14(12):1985-93. doi: 10.1111/pme.12255. Epub 2013 Oct 9. PMID 24119077
- [Background] Robinson-Papp J, Sharma S, Dhadwal N, Simpson DM, Morgello S. Optimizing measures of HIV-associated neuropathy. Muscle Nerve. 2015 Jan;51(1):56-64. doi: 10.1002/mus.24282. Epub 2014 Nov 21. PMID 24809943
- [Background] Chou R, Turner JA, Devine EB, Hansen RN, Sullivan SD, Blazina I, Dana T, Bougatsos C, Deyo RA. The effectiveness and risks of long-term opioid therapy for chronic pain: a systematic review for a National Institutes of Health Pathways to Prevention Workshop. Ann Intern Med. 2015 Feb 17;162(4):276-86. doi: 10.7326/M14-2559. PMID 25581257
- [Background] Liu B, Liu X, Tang SJ. Interactions of Opioids and HIV Infection in the Pathogenesis of Chronic Pain. Front Microbiol. 2016 Feb 10;7:103. doi: 10.3389/fmicb.2016.00103. eCollection 2016. PMID 26903982
- [Background] Gandhi RT, McMahon DK, Bosch RJ, Lalama CM, Cyktor JC, Macatangay BJ, Rinaldo CR, Riddler SA, Hogg E, Godfrey C, Collier AC, Eron JJ, Mellors JW; ACTG A5321 Team. Levels of HIV-1 persistence on antiretroviral therapy are not associated with markers of inflammation or activation. PLoS Pathog. 2017 Apr 20;13(4):e1006285. doi: 10.1371/journal.ppat.1006285. eCollection 2017 Apr. PMID 28426825
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain - United States, 2016. MMWR Recomm Rep. 2016 Mar 18;65(1):1-49. doi: 10.15585/mmwr.rr6501e1. PMID 26987082
- [Background] Vervest ACM, Schimmel GH. Taxonomy of pain of the IASP. Pain. 1988 Sep;34(3):318-321. doi: 10.1016/0304-3959(88)90129-7. No abstract available. PMID 3054730
- [Background] Turk DC, Wilson HD, Cahana A. Treatment of chronic non-cancer pain. Lancet. 2011 Jun 25;377(9784):2226-35. doi: 10.1016/S0140-6736(11)60402-9. PMID 21704872
- [Background] Jiao JM, So E, Jebakumar J, George MC, Simpson DM, Robinson-Papp J. Chronic pain disorders in HIV primary care: clinical characteristics and association with healthcare utilization. Pain. 2016 Apr;157(4):931-937. doi: 10.1097/j.pain.0000000000000462. PMID 26683238
- [Background] Robinson-Papp J, Morgello S, Vaida F, Fitzsimons C, Simpson DM, Elliott KJ, Al-Lozi M, Gelman BB, Clifford D, Marra CM, McCutchan JA, Atkinson JH, Dworkin RH, Grant I, Ellis R. Association of self-reported painful symptoms with clinical and neurophysiologic signs in HIV-associated sensory neuropathy. Pain. 2010 Dec;151(3):732-736. doi: 10.1016/j.pain.2010.08.045. Epub 2010 Sep 20. PMID 20851521
- [Background] Morgello S, Estanislao L, Simpson D, Geraci A, DiRocco A, Gerits P, Ryan E, Yakoushina T, Khan S, Mahboob R, Naseer M, Dorfman D, Sharp V; Manhattan HIV Brain Bank. HIV-associated distal sensory polyneuropathy in the era of highly active antiretroviral therapy: the Manhattan HIV Brain Bank. Arch Neurol. 2004 Apr;61(4):546-51. doi: 10.1001/archneur.61.4.546. PMID 15096404
- [Background] Ellis RJ, Rosario D, Clifford DB, McArthur JC, Simpson D, Alexander T, Gelman BB, Vaida F, Collier A, Marra CM, Ances B, Atkinson JH, Dworkin RH, Morgello S, Grant I; CHARTER Study Group. Continued high prevalence and adverse clinical impact of human immunodeficiency virus-associated sensory neuropathy in the era of combination antiretroviral therapy: the CHARTER Study. Arch Neurol. 2010 May;67(5):552-8. doi: 10.1001/archneurol.2010.76. PMID 20457954
- [Background] Lehmann HC, Chen W, Borzan J, Mankowski JL, Hoke A. Mitochondrial dysfunction in distal axons contributes to human immunodeficiency virus sensory neuropathy. Ann Neurol. 2011 Jan;69(1):100-10. doi: 10.1002/ana.22150. Epub 2010 Nov 8. PMID 21280080
- [Background] Malvar J, Vaida F, Sanders CF, Atkinson JH, Bohannon W, Keltner J, Robinson-Papp J, Simpson DM, Marra CM, Clifford DB, Gelman B, Fan J, Grant I, Ellis RJ; CHARTER Group. Predictors of new-onset distal neuropathic pain in HIV-infected individuals in the era of combination antiretroviral therapy. Pain. 2015 Apr;156(4):731-739. doi: 10.1097/01.j.pain.0000461252.75089.bf. PMID 25659067
- [Background] Levy B, Paulozzi L, Mack KA, Jones CM. Trends in Opioid Analgesic-Prescribing Rates by Specialty, U.S., 2007-2012. Am J Prev Med. 2015 Sep;49(3):409-13. doi: 10.1016/j.amepre.2015.02.020. Epub 2015 Apr 18. PMID 25896191
- [Background] Silverberg MJ, Ray GT, Saunders K, Rutter CM, Campbell CI, Merrill JO, Sullivan MD, Banta-Green CJ, Von Korff M, Weisner C. Prescription long-term opioid use in HIV-infected patients. Clin J Pain. 2012 Jan;28(1):39-46. doi: 10.1097/AJP.0b013e3182201a0f. PMID 21677568
- [Background] Edelman EJ, Gordon K, Becker WC, Goulet JL, Skanderson M, Gaither JR, Brennan Braden J, Gordon AJ, Kerns RD, Justice AC, Fiellin DA. Receipt of opioid analgesics by HIV-infected and uninfected patients. J Gen Intern Med. 2013 Jan;28(1):82-90. doi: 10.1007/s11606-012-2189-z. Epub 2012 Aug 16. PMID 22895747
- [Background] Merlin JS, Tamhane A, Starrels JL, Kertesz S, Saag M, Cropsey K. Factors Associated with Prescription of Opioids and Co-prescription of Sedating Medications in Individuals with HIV. AIDS Behav. 2016 Mar;20(3):687-98. doi: 10.1007/s10461-015-1178-8. PMID 26487298
- [Background] Frenk SM, Porter KS, Paulozzi LJ. Prescription opioid analgesic use among adults: United States, 1999-2012. NCHS Data Brief. 2015 Feb;(189):1-8. PMID 25714043
- [Background] Merlin JS, Long D, Becker WC, Cachay ER, Christopoulos KA, Claborn K, Crane HM, Edelman EJ, Harding R, Kertesz SG, Liebschutz JM, Mathews WC, Mugavero MJ, Napravnik S, C O'Cleirigh C, Saag MS, Starrels JL, Gross R. Brief Report: The Association of Chronic Pain and Long-Term Opioid Therapy With HIV Treatment Outcomes. J Acquir Immune Defic Syndr. 2018 Sep 1;79(1):77-82. doi: 10.1097/QAI.0000000000001741. PMID 29771793
- [Background] Noble M, Treadwell JR, Tregear SJ, Coates VH, Wiffen PJ, Akafomo C, Schoelles KM. Long-term opioid management for chronic noncancer pain. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD006605. doi: 10.1002/14651858.CD006605.pub2. PMID 20091598
- [Background] Koeppe J, Armon C, Lyda K, Nielsen C, Johnson S. Ongoing pain despite aggressive opioid pain management among persons with HIV. Clin J Pain. 2010 Mar-Apr;26(3):190-8. doi: 10.1097/AJP.0b013e3181b91624. PMID 20173432
- [Background] Solomon DH, Rassen JA, Glynn RJ, Garneau K, Levin R, Lee J, Schneeweiss S. The comparative safety of opioids for nonmalignant pain in older adults. Arch Intern Med. 2010 Dec 13;170(22):1979-86. doi: 10.1001/archinternmed.2010.450. PMID 21149754
- [Background] Li L, Setoguchi S, Cabral H, Jick S. Opioid use for noncancer pain and risk of myocardial infarction amongst adults. J Intern Med. 2013 May;273(5):511-26. doi: 10.1111/joim.12035. Epub 2013 Feb 16. PMID 23331508
- [Background] Li L, Setoguchi S, Cabral H, Jick S. Opioid use for noncancer pain and risk of fracture in adults: a nested case-control study using the general practice research database. Am J Epidemiol. 2013 Aug 15;178(4):559-69. doi: 10.1093/aje/kwt013. Epub 2013 May 2. PMID 23639937
- [Background] Reddy RG, Aung T, Karavitaki N, Wass JA. Opioid induced hypogonadism. BMJ. 2010 Aug 31;341:c4462. doi: 10.1136/bmj.c4462. PMID 20807731
- [Background] Dunn KM, Saunders KW, Rutter CM, Banta-Green CJ, Merrill JO, Sullivan MD, Weisner CM, Silverberg MJ, Campbell CI, Psaty BM, Von Korff M. Opioid prescriptions for chronic pain and overdose: a cohort study. Ann Intern Med. 2010 Jan 19;152(2):85-92. doi: 10.7326/0003-4819-152-2-201001190-00006. PMID 20083827
- [Background] Morasco BJ, Dobscha SK. Prescription medication misuse and substance use disorder in VA primary care patients with chronic pain. Gen Hosp Psychiatry. 2008 Mar-Apr;30(2):93-9. doi: 10.1016/j.genhosppsych.2007.12.004. PMID 18291290
- [Background] Bohnert AS, Valenstein M, Bair MJ, Ganoczy D, McCarthy JF, Ilgen MA, Blow FC. Association between opioid prescribing patterns and opioid overdose-related deaths. JAMA. 2011 Apr 6;305(13):1315-21. doi: 10.1001/jama.2011.370. PMID 21467284
- [Background] Gomes T, Mamdani MM, Dhalla IA, Paterson JM, Juurlink DN. Opioid dose and drug-related mortality in patients with nonmalignant pain. Arch Intern Med. 2011 Apr 11;171(7):686-91. doi: 10.1001/archinternmed.2011.117. PMID 21482846
- [Background] Paulozzi LJ, Kilbourne EM, Shah NG, Nolte KB, Desai HA, Landen MG, Harvey W, Loring LD. A history of being prescribed controlled substances and risk of drug overdose death. Pain Med. 2012 Jan;13(1):87-95. doi: 10.1111/j.1526-4637.2011.01260.x. Epub 2011 Oct 25. PMID 22026451
- [Background] Webster LR, Cochella S, Dasgupta N, Fakata KL, Fine PG, Fishman SM, Grey T, Johnson EM, Lee LK, Passik SD, Peppin J, Porucznik CA, Ray A, Schnoll SH, Stieg RL, Wakeland W. An analysis of the root causes for opioid-related overdose deaths in the United States. Pain Med. 2011 Jun;12 Suppl 2:S26-35. doi: 10.1111/j.1526-4637.2011.01134.x. PMID 21668754
- [Background] Weisberg DF, Gordon KS, Barry DT, Becker WC, Crystal S, Edelman EJ, Gaither J, Gordon AJ, Goulet J, Kerns RD, Moore BA, Tate J, Justice AC, Fiellin DA. Long-term Prescription of Opioids and/or Benzodiazepines and Mortality Among HIV-Infected and Uninfected Patients. J Acquir Immune Defic Syndr. 2015 Jun 1;69(2):223-33. doi: 10.1097/QAI.0000000000000591. PMID 26009831
- [Background] Merlin JS, Young SR, Starrels JL, Azari S, Edelman EJ, Pomeranz J, Roy P, Saini S, Becker WC, Liebschutz JM. Managing Concerning Behaviors in Patients Prescribed Opioids for Chronic Pain: A Delphi Study. J Gen Intern Med. 2018 Feb;33(2):166-176. doi: 10.1007/s11606-017-4211-y. Epub 2017 Dec 4. PMID 29204977
- [Background] Scherrer JF, Svrakic DM, Freedland KE, Chrusciel T, Balasubramanian S, Bucholz KK, Lawler EV, Lustman PJ. Prescription opioid analgesics increase the risk of depression. J Gen Intern Med. 2014 Mar;29(3):491-9. doi: 10.1007/s11606-013-2648-1. Epub 2013 Oct 29. PMID 24165926
- [Background] Smallwood N, Politis J, Le B. Prescription opioid use in advanced COPD: benefits, perils and controversies. Eur Respir J. 2017 Jun 22;49(6):1700690. doi: 10.1183/13993003.00690-2017. Print 2017 Jun. No abstract available. PMID 28642317
- [Background] El-Hage N, Gurwell JA, Singh IN, Knapp PE, Nath A, Hauser KF. Synergistic increases in intracellular Ca2+, and the release of MCP-1, RANTES, and IL-6 by astrocytes treated with opiates and HIV-1 Tat. Glia. 2005 Apr 15;50(2):91-106. doi: 10.1002/glia.20148. PMID 15630704
- [Background] Yu Y, Huang X, Di Y, Qu L, Fan N. Effect of CXCL12/CXCR4 signaling on neuropathic pain after chronic compression of dorsal root ganglion. Sci Rep. 2017 Jul 18;7(1):5707. doi: 10.1038/s41598-017-05954-1. PMID 28720830
- [Background] Wilson NM, Jung H, Ripsch MS, Miller RJ, White FA. CXCR4 signaling mediates morphine-induced tactile hyperalgesia. Brain Behav Immun. 2011 Mar;25(3):565-73. doi: 10.1016/j.bbi.2010.12.014. Epub 2010 Dec 28. PMID 21193025
- [Background] Davey RT Jr, Bhat N, Yoder C, Chun TW, Metcalf JA, Dewar R, Natarajan V, Lempicki RA, Adelsberger JW, Miller KD, Kovacs JA, Polis MA, Walker RE, Falloon J, Masur H, Gee D, Baseler M, Dimitrov DS, Fauci AS, Lane HC. HIV-1 and T cell dynamics after interruption of highly active antiretroviral therapy (HAART) in patients with a history of sustained viral suppression. Proc Natl Acad Sci U S A. 1999 Dec 21;96(26):15109-14. doi: 10.1073/pnas.96.26.15109. PMID 10611346
- [Background] Deeks S. Towards an HIV cure. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19479. doi: 10.7448/IAS.17.4.19479. eCollection 2014. PMID 25393988
- [Background] Chun TW, Stuyver L, Mizell SB, Ehler LA, Mican JA, Baseler M, Lloyd AL, Nowak MA, Fauci AS. Presence of an inducible HIV-1 latent reservoir during highly active antiretroviral therapy. Proc Natl Acad Sci U S A. 1997 Nov 25;94(24):13193-7. doi: 10.1073/pnas.94.24.13193. PMID 9371822
- [Background] Finzi D, Hermankova M, Pierson T, Carruth LM, Buck C, Chaisson RE, Quinn TC, Chadwick K, Margolick J, Brookmeyer R, Gallant J, Markowitz M, Ho DD, Richman DD, Siliciano RF. Identification of a reservoir for HIV-1 in patients on highly active antiretroviral therapy. Science. 1997 Nov 14;278(5341):1295-300. doi: 10.1126/science.278.5341.1295. PMID 9360927
- [Background] Wong JK, Hezareh M, Gunthard HF, Havlir DV, Ignacio CC, Spina CA, Richman DD. Recovery of replication-competent HIV despite prolonged suppression of plasma viremia. Science. 1997 Nov 14;278(5341):1291-5. doi: 10.1126/science.278.5341.1291. PMID 9360926
- [Background] Siliciano JM, Siliciano RF. The Remarkable Stability of the Latent Reservoir for HIV-1 in Resting Memory CD4+ T Cells. J Infect Dis. 2015 Nov 1;212(9):1345-7. doi: 10.1093/infdis/jiv219. Epub 2015 Apr 15. No abstract available. PMID 25877551
- [Background] Zhang JM, An J. Cytokines, inflammation, and pain. Int Anesthesiol Clin. 2007 Spring;45(2):27-37. doi: 10.1097/AIA.0b013e318034194e. PMID 17426506
- [Background] Backonja MM, Attal N, Baron R, Bouhassira D, Drangholt M, Dyck PJ, Edwards RR, Freeman R, Gracely R, Haanpaa MH, Hansson P, Hatem SM, Krumova EK, Jensen TS, Maier C, Mick G, Rice AS, Rolke R, Treede RD, Serra J, Toelle T, Tugnoli V, Walk D, Walalce MS, Ware M, Yarnitsky D, Ziegler D. Value of quantitative sensory testing in neurological and pain disorders: NeuPSIG consensus. Pain. 2013 Sep;154(9):1807-1819. doi: 10.1016/j.pain.2013.05.047. Epub 2013 Jun 3. PMID 23742795
- [Background] Cruz-Almeida Y, Fillingim RB. Can quantitative sensory testing move us closer to mechanism-based pain management? Pain Med. 2014 Jan;15(1):61-72. doi: 10.1111/pme.12230. Epub 2013 Sep 6. PMID 24010588
- [Background] Goodin BR, Bulls HW, Herbert MS, Schmidt J, King CD, Glover TL, Sotolongo A, Sibille KT, Cruz-Almeida Y, Staud R, Fessler BJ, Redden DT, Bradley LA, Fillingim RB. Temporal summation of pain as a prospective predictor of clinical pain severity in adults aged 45 years and older with knee osteoarthritis: ethnic differences. Psychosom Med. 2014 May;76(4):302-10. doi: 10.1097/PSY.0000000000000058. PMID 24804882
- [Background] Stringer EA, Baker KS, Carroll IR, Montoya JG, Chu L, Maecker HT, Younger JW. Daily cytokine fluctuations, driven by leptin, are associated with fatigue severity in chronic fatigue syndrome: evidence of inflammatory pathology. J Transl Med. 2013 Apr 9;11:93. doi: 10.1186/1479-5876-11-93. PMID 23570606
- [Background] Parkitny L, Middleton S, Baker K, Younger J. Evidence for abnormal cytokine expression in Gulf War Illness: A preliminary analysis of daily immune monitoring data. BMC Immunol. 2015 Sep 30;16:57. doi: 10.1186/s12865-015-0122-z. PMID 26420016
- [Background] Younger J, Kapphahn K, Brennan K, Sullivan SD, Stefanick ML. Association of Leptin with Body Pain in Women. J Womens Health (Larchmt). 2016 Jul;25(7):752-60. doi: 10.1089/jwh.2015.5509. Epub 2016 Mar 30. PMID 27028709
- [Background] Merlin JS, Westfall AO, Heath SL, Goodin BR, Stewart JC, Sorge RE, Younger J. Brief Report: IL-1beta Levels Are Associated With Chronic Multisite Pain in People Living With HIV. J Acquir Immune Defic Syndr. 2017 Aug 1;75(4):e99-e103. doi: 10.1097/QAI.0000000000001377. PMID 28328552
- [Background] Merlin JS, Westfall AO, Chamot E, Saag M, Walcott M, Ritchie C, Kertesz S. Quantitative Evaluation of an Instrument to Identify Chronic Pain in HIV-Infected Individuals. AIDS Res Hum Retroviruses. 2015 Jun;31(6):623-7. doi: 10.1089/AID.2014.0362. Epub 2015 Mar 12. PMID 25693683
- [Background] Goodin BR, Owens MA, Yessick LR, Rainey RL, Okunbor JI, White DM, Mushatt KA, Harmon OA, Heath SL, Merlin JS. Detectable Viral Load May Be Associated with Increased Pain Sensitivity in Persons Living with HIV: Preliminary Findings. Pain Med. 2017 Dec 1;18(12):2289-2295. doi: 10.1093/pm/pnx057. PMID 28398572
- [Background] England JD, Gronseth GS, Franklin G, Miller RG, Asbury AK, Carter GT, Cohen JA, Fisher MA, Howard JF, Kinsella LJ, Latov N, Lewis RA, Low PA, Sumner AJ; American Academy of Neurology; American Association of Electrodiagnostic Medicine; American Academy of Physical Medicine and Rehabilitation. Distal symmetric polyneuropathy: a definition for clinical research: report of the American Academy of Neurology, the American Association of Electrodiagnostic Medicine, and the American Academy of Physical Medicine and Rehabilitation. Neurology. 2005 Jan 25;64(2):199-207. doi: 10.1212/01.WNL.0000149522.32823.EA. PMID 15668414
- [Background] Robinson-Papp J, Gonzalez-Duarte A, Simpson DM, Rivera-Mindt M, Morgello S; Manhattan HIV Brain Bank. The roles of ethnicity and antiretrovirals in HIV-associated polyneuropathy: a pilot study. J Acquir Immune Defic Syndr. 2009 Aug 15;51(5):569-73. doi: 10.1097/QAI.0b013e3181adcefa. PMID 19521250
- [Background] Robinson-Papp J, Gelman BB, Grant I, Singer E, Gensler G, Morgello S; National NeuroAIDS Tissue Consortium. Substance abuse increases the risk of neuropathy in an HIV-infected cohort. Muscle Nerve. 2012 Apr;45(4):471-6. doi: 10.1002/mus.23231. PMID 22431078
- [Background] Simpson DM, Robinson-Papp J, Van J, Stoker M, Jacobs H, Snijder RJ, Schregardus DS, Long SK, Lambourg B, Katz N. Capsaicin 8% Patch in Painful Diabetic Peripheral Neuropathy: A Randomized, Double-Blind, Placebo-Controlled Study. J Pain. 2017 Jan;18(1):42-53. doi: 10.1016/j.jpain.2016.09.008. Epub 2016 Oct 13. PMID 27746370
- [Background] Samikkannu T, Rao KV, Arias AY, Kalaichezian A, Sagar V, Yoo C, Nair MP. HIV infection and drugs of abuse: role of acute phase proteins. J Neuroinflammation. 2013 Sep 17;10:113. doi: 10.1186/1742-2094-10-113. PMID 24044608
- [Background] Schomberg D, Ahmed M, Miranpuri G, Olson J, Resnick DK. Neuropathic pain: role of inflammation, immune response, and ion channel activity in central injury mechanisms. Ann Neurosci. 2012 Jul;19(3):125-32. doi: 10.5214/ans.0972.7531.190309. PMID 25205985
- [Background] Zhao H, Alam A, Chen Q, A Eusman M, Pal A, Eguchi S, Wu L, Ma D. The role of microglia in the pathobiology of neuropathic pain development: what do we know? Br J Anaesth. 2017 Apr 1;118(4):504-516. doi: 10.1093/bja/aex006. PMID 28403399
- [Background] Sun C, Zhang J, Chen L, Liu T, Xu G, Li C, Yuan W, Xu H, Su Z. IL-17 contributed to the neuropathic pain following peripheral nerve injury by promoting astrocyte proliferation and secretion of proinflammatory cytokines. Mol Med Rep. 2017 Jan;15(1):89-96. doi: 10.3892/mmr.2016.6018. Epub 2016 Dec 9. PMID 27959414
- [Background] Clark AK, Old EA, Malcangio M. Neuropathic pain and cytokines: current perspectives. J Pain Res. 2013 Nov 21;6:803-14. doi: 10.2147/JPR.S53660. eCollection 2013. PMID 24294006
- [Background] Zheng L, Bosch RJ, Chan ES, Read S, Kearney M, Margolis DM, Mellors JW, Eron JJ, Gandhi RT; DS Clinical Trials Group (ACTG) A5244 Team. Predictors of residual viraemia in patients on long-term suppressive antiretroviral therapy. Antivir Ther. 2013;18(1):39-43. doi: 10.3851/IMP2323. Epub 2012 Aug 22. PMID 22914318
- [Background] Riddler SA, Aga E, Bosch RJ, Bastow B, Bedison M, Vagratian D, Vaida F, Eron JJ, Gandhi RT, Mellors JW; ACTG A5276s Protocol Team. Continued Slow Decay of the Residual Plasma Viremia Level in HIV-1-Infected Adults Receiving Long-term Antiretroviral Therapy. J Infect Dis. 2016 Feb 15;213(4):556-60. doi: 10.1093/infdis/jiv433. Epub 2015 Sep 2. PMID 26333941
- [Background] Cillo AR, Vagratian D, Bedison MA, Anderson EM, Kearney MF, Fyne E, Koontz D, Coffin JM, Piatak M Jr, Mellors JW. Improved single-copy assays for quantification of persistent HIV-1 viremia in patients on suppressive antiretroviral therapy. J Clin Microbiol. 2014 Nov;52(11):3944-51. doi: 10.1128/JCM.02060-14. Epub 2014 Sep 3. PMID 25187636
- [Background] Cillo AR, Sobolewski MD, Bosch RJ, Fyne E, Piatak M Jr, Coffin JM, Mellors JW. Quantification of HIV-1 latency reversal in resting CD4+ T cells from patients on suppressive antiretroviral therapy. Proc Natl Acad Sci U S A. 2014 May 13;111(19):7078-83. doi: 10.1073/pnas.1402873111. Epub 2014 Mar 31. PMID 24706775
- [Background] Palmer S, Wiegand AP, Maldarelli F, Bazmi H, Mican JM, Polis M, Dewar RL, Planta A, Liu S, Metcalf JA, Mellors JW, Coffin JM. New real-time reverse transcriptase-initiated PCR assay with single-copy sensitivity for human immunodeficiency virus type 1 RNA in plasma. J Clin Microbiol. 2003 Oct;41(10):4531-6. doi: 10.1128/JCM.41.10.4531-4536.2003. PMID 14532178
- [Background] Ho YC, Shan L, Hosmane NN, Wang J, Laskey SB, Rosenbloom DI, Lai J, Blankson JN, Siliciano JD, Siliciano RF. Replication-competent noninduced proviruses in the latent reservoir increase barrier to HIV-1 cure. Cell. 2013 Oct 24;155(3):540-51. doi: 10.1016/j.cell.2013.09.020. Epub 2013 Oct 24. PMID 24243014
- [Background] Pollack RA, Jones RB, Pertea M, Bruner KM, Martin AR, Thomas AS, Capoferri AA, Beg SA, Huang SH, Karandish S, Hao H, Halper-Stromberg E, Yong PC, Kovacs C, Benko E, Siliciano RF, Ho YC. Defective HIV-1 Proviruses Are Expressed and Can Be Recognized by Cytotoxic T Lymphocytes, which Shape the Proviral Landscape. Cell Host Microbe. 2017 Apr 12;21(4):494-506.e4. doi: 10.1016/j.chom.2017.03.008. PMID 28407485
- [Background] Bui JK, Mellors JW, Cillo AR. HIV-1 Virion Production from Single Inducible Proviruses following T-Cell Activation Ex Vivo. J Virol. 2015 Nov 11;90(3):1673-6. doi: 10.1128/JVI.02520-15. Print 2016 Feb 1. PMID 26559835
- [Background] Hong F, Aga E, Cillo AR, Yates AL, Besson G, Fyne E, Koontz DL, Jennings C, Zheng L, Mellors JW. Novel Assays for Measurement of Total Cell-Associated HIV-1 DNA and RNA. J Clin Microbiol. 2016 Apr;54(4):902-11. doi: 10.1128/JCM.02904-15. Epub 2016 Jan 13. PMID 26763968
- [Background] Marchetti G, Tincati C, Silvestri G. Microbial translocation in the pathogenesis of HIV infection and AIDS. Clin Microbiol Rev. 2013 Jan;26(1):2-18. doi: 10.1128/CMR.00050-12. PMID 23297256
- [Background] Caradonna L, Amati L, Magrone T, Pellegrino NM, Jirillo E, Caccavo D. Enteric bacteria, lipopolysaccharides and related cytokines in inflammatory bowel disease: biological and clinical significance. J Endotoxin Res. 2000;6(3):205-14. PMID 11052175
- [Background] Caliendo AM, St George K, Allega J, Bullotta AC, Gilbane L, Rinaldo CR. Distinguishing cytomegalovirus (CMV) infection and disease with CMV nucleic acid assays. J Clin Microbiol. 2002 May;40(5):1581-6. doi: 10.1128/JCM.40.5.1581-1586.2002. PMID 11980925
- [Background] Martin A, Rief W, Klaiberg A, Braehler E. Validity of the Brief Patient Health Questionnaire Mood Scale (PHQ-9) in the general population. Gen Hosp Psychiatry. 2006 Jan-Feb;28(1):71-7. doi: 10.1016/j.genhosppsych.2005.07.003. PMID 16377369
- [Background] Newcombe DA, Humeniuk RE, Ali R. Validation of the World Health Organization Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): report of results from the Australian site. Drug Alcohol Rev. 2005 May;24(3):217-26. doi: 10.1080/09595230500170266. PMID 16096125
- [Background] Dworkin RH, Turk DC, Wyrwich KW, Beaton D, Cleeland CS, Farrar JT, Haythornthwaite JA, Jensen MP, Kerns RD, Ader DN, Brandenburg N, Burke LB, Cella D, Chandler J, Cowan P, Dimitrova R, Dionne R, Hertz S, Jadad AR, Katz NP, Kehlet H, Kramer LD, Manning DC, McCormick C, McDermott MP, McQuay HJ, Patel S, Porter L, Quessy S, Rappaport BA, Rauschkolb C, Revicki DA, Rothman M, Schmader KE, Stacey BR, Stauffer JW, von Stein T, White RE, Witter J, Zavisic S. Interpreting the clinical importance of treatment outcomes in chronic pain clinical trials: IMMPACT recommendations. J Pain. 2008 Feb;9(2):105-21. doi: 10.1016/j.jpain.2007.09.005. Epub 2007 Dec 11. PMID 18055266
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Doyle HH, Murphy AZ. Sex differences in innate immunity and its impact on opioid pharmacology. J Neurosci Res. 2017 Jan 2;95(1-2):487-499. doi: 10.1002/jnr.23852. PMID 27870418
- [Background] Wegner A, Benson S, Rebernik L, Spreitzer I, Jager M, Schedlowski M, Elsenbruch S, Engler H. Sex differences in the pro-inflammatory cytokine response to endotoxin unfold in vivo but not ex vivo in healthy humans. Innate Immun. 2017 Jul;23(5):432-439. doi: 10.1177/1753425917707026. Epub 2017 Apr 26. PMID 28443392
- [Background] Sorge RE, Totsch SK. Sex Differences in Pain. J Neurosci Res. 2017 Jun;95(6):1271-1281. doi: 10.1002/jnr.23841. Epub 2016 Jul 25. PMID 27452349
- [Background] Melchior M, Poisbeau P, Gaumond I, Marchand S. Insights into the mechanisms and the emergence of sex-differences in pain. Neuroscience. 2016 Dec 3;338:63-80. doi: 10.1016/j.neuroscience.2016.05.007. Epub 2016 May 12. PMID 27180284
- [Background] Frank JW, Lovejoy TI, Becker WC, Morasco BJ, Koenig CJ, Hoffecker L, Dischinger HR, Dobscha SK, Krebs EE. Patient Outcomes in Dose Reduction or Discontinuation of Long-Term Opioid Therapy: A Systematic Review. Ann Intern Med. 2017 Aug 1;167(3):181-191. doi: 10.7326/M17-0598. Epub 2017 Jul 11. PMID 28715848
- [Derived] McGill LS, Clay OJ, Edwards KA, Jones KF, Long DM, Johnson MO, Bair MJ, Browne LE, Liebschutz JM, Demonte W, Agil D, Burkholder G, Durr AL, Farel CE, Johnson B, Orris SM, Napravnik S, Thomas T, Merlin JS. Trajectories of Pain Impact and Pain Self-Efficacy in People With HIV and Chronic Pain: Extending Findings From the Skills TO Manage Pain Randomized Clinical Trial. J Acquir Immune Defic Syndr. 2025 Dec 1;100(4):347-354. doi: 10.1097/QAI.0000000000003739. PMID 40748350
- [Derived] Edwards KA, Long D, Jones KF, Durr AL, Farel CE, Liebschutz JM, Bair MJ, Agil D, Napravnik S, Browne L, Johnson B, Thomas T, Burkholder G, Clay OJ, Demonte W, Orris SM, Johnson MO, Merlin J. The Skills to Manage Pain Randomized Trial: Results of Antiretroviral Therapy Adherence, HIV Primary Care Retention, and Virologic Suppression Outcomes. J Acquir Immune Defic Syndr. 2025 Oct 1;100(2):180-185. doi: 10.1097/QAI.0000000000003706. PMID 40530923
- [Derived] Edwards KA, Smith KJ, Jones KF, Bair MJ, Liebschutz JM, McGill LS, Agil D, Johnson MO, Thomas T, Clay OJ, Farel CE, Napravnik S, Long D, Burkholder G, Browne L, Durr AL, Johnson B, Demonte W, Orris SM, Merlin JS. Cost-Effectiveness of a Tailored Pain Self-Management Intervention Compared With Enhanced Usual Care Among People With HIV and Chronic Pain: An Economic Evaluation. J Acquir Immune Defic Syndr. 2025 Aug 1;99(4):341-348. doi: 10.1097/QAI.0000000000003671. PMID 40179206
- [Derived] Jones KF, Long DM, Bair MJ, Agil D, Browne L, Burkholder G, Clay OJ, Conder K, Durr AL, Farel CE, King K, Johnson B, Liebschutz JM, Demonte W, Leone M, Mullen L, Orris SM, Thomas T, Johnson M, Napravnik S, Merlin JS. Efficacy of a Pain Self-Management Intervention Tailored to People With HIV: A Randomized Clinical Trial. JAMA Intern Med. 2024 Sep 1;184(9):1074-1082. doi: 10.1001/jamainternmed.2024.3071. PMID 39008317
- [Derived] Jones KF, Bair MJ, Orris SM, Johnson M, Liebschutz JM, Demonte W, Clay OJ, Durr AL, Farel CE, Agil D, Burkholder G, Johnson B, Conder K, Leone M, Napravnik S, Thomas T, Browne L, King K, Mullen L, Merlin J. Evaluation of the efficacy and mechanisms of a novel intervention for chronic pain tailored to people with HIV: The STOMP protocol. Contemp Clin Trials. 2023 Jun;129:107163. doi: 10.1016/j.cct.2023.107163. Epub 2023 Mar 21. PMID 36958702

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Skills to Manage Pain (STOMP) | Comparison Group
Started | 139 | 139
Completed | 136 | 139
Not Completed | 3 | 0
Not completed — Found to be ineligible postrandomization | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Skills to Manage Pain (STOMP) | Comparison Group | Total
Number analyzed (Participants) | 139 | 139 | 278
Age, Customized [Mean (Standard Deviation); unit: years] | 53.7 (9.6) | 53.3 (10.4) | 53.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 65 | 132
  Male | 72 | 74 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 137 | 138 | 275
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 107 | 118 | 225
  White | 27 | 19 | 46
  Other or American Indian/Alaska Native | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 139 | 139 | 278
Site [Count of Participants; unit: Participants]
  University of Alabama at Birmingham | 67 | 72 | 139
  University of North Carolina-Chapel Hill | 72 | 67 | 139
Detectable viral load, >200 copies/mL [Count of Participants; unit: Participants]
  No | 120 | 116 | 236
  Yes | 6 | 8 | 14
  Unknown | 13 | 15 | 28
Currently taking any anti-HIV medications [Count of Participants; unit: Participants]
  No | 4 | 2 | 6
  Yes | 135 | 136 | 271
  Unknown | 0 | 1 | 1
Brief Pain Inventory (BPI) Total Score [Mean (Standard Deviation); unit: units on a scale] — The Brief Pain Inventory measures pain severity and impact on daily functioning. Includes 4 items assessing pain severity (worst/least/average/current) and 7 items assessing pain interference with general activity, mood, walking, work, relations with others, sleep, and life enjoyment. Each item and measure is rated from 0-10 with higher scores indicating worse pain severity and greater pain interference. The Pain Severity Subscore is the average of 4 severity items, the Functional Interference Subscore is the average of 7 interference items, and the Total Score is the average of all 11 items.
  units on a scale | 6.3 (1.7) | 6.4 (1.7) | 6.4 (1.7)
Brief Pain Inventory (BPI) Pain Severity Subscore [Mean (Standard Deviation); unit: units on a scale] — The Brief Pain Inventory measures pain severity and impact on daily functioning. Includes 4 items assessing pain severity (worst/least/average/current) and 7 items assessing pain interference with general activity, mood, walking, work, relations with others, sleep, and life enjoyment. Each item and measure is rated from 0-10 with higher scores indicating worse pain severity and greater pain interference. The Pain Severity Subscore is the average of 4 severity items, the Functional Interference Subscore is the average of 7 interference items, and the Total Score is the average of all 11 items.
  units on a scale | 6.4 (1.8) | 6.6 (1.8) | 6.5 (1.8)
Brief Pain Inventory (BPI) Functional Interference Subscore [Mean (Standard Deviation); unit: units on a scale] — The Brief Pain Inventory measures pain severity and impact on daily functioning. Includes 4 items assessing pain severity (worst/least/average/current) and 7 items assessing pain interference with general activity, mood, walking, work, relations with others, sleep, and life enjoyment. Each item and measure is rated from 0-10 with higher scores indicating worse pain severity and greater pain interference. The Pain Severity Subscore is the average of 4 severity items, the Functional Interference Subscore is the average of 7 interference items, and the Total Score is the average of all 11 items.
  units on a scale | 6.5 (2.2) | 6.4 (2.3) | 6.4 (2.2)
Taken an opioid or narcotic for pain for 3 months or more [Count of Participants; unit: Participants]
  No | 106 | 107 | 213
  Yes | 33 | 32 | 65
Multisite pain (>3 sites of pain) [Count of Participants; unit: Participants]
  No | 32 | 30 | 62
  Yes | 107 | 109 | 216
Pain locations [Count of Participants; unit: Participants]
  Numbness or tingling in hands and/or feet | 75 | 71 | 146
  Headache | 39 | 43 | 82
  Abdominal | 31 | 30 | 61
  Lower back | 109 | 101 | 210
  Hip | 64 | 67 | 131
  Shoulder | 64 | 57 | 121
  Knee | 75 | 75 | 150
  Pain everywhere in the body | 28 | 28 | 56
  Other | 65 | 70 | 135
Cocaine use history [Count of Participants; unit: Participants]
  None | 69 | 58 | 127
  Past use | 66 | 78 | 144
  Current use | 4 | 2 | 6
  Unknown | 0 | 1 | 1
The Pain, Enjoyment and General Activity (PEG) scale [Mean (Standard Deviation); unit: units on a scale] — The Pain, Enjoyment and General Activity (PEG) scale measures pain severity and enjoyment of activities with scores ranging from 0 to 10. Higher scores indicate worse pain and greater interference with daily activities. The total score is the average of 3 items assessing pain intensity, enjoyment of life, and general activity.
  units on a scale | 7.4 (1.6) | 7.5 (1.7) | 7.5 (1.6)
The Pain Self-Efficacy Questionnaire (PSEQ) [Mean (Standard Deviation); unit: units on a scale] — The Pain Self-Efficacy Questionnaire (PSEQ) assesses an individual's confidence in their ability to perform daily activities despite pain. The total score is the sum of 10 items, each rated from 0 to 6, resulting in a range of 0 to 60. Higher scores indicate greater self-efficacy and a stronger belief in one's ability to manage daily tasks while experiencing pain.
  units on a scale | 34.6 (13.4) | 32.5 (15.4) | 33.6 (14.5)
The Patient Health Questionnaire-8 (PHQ-8) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-8 (PHQ-8) is an 8-item self-report measure assessing depressive symptoms over the past two weeks. Each item is rated from 0 to 3, with the total score (0-24) calculated by adding all responses, with higher scores indicating more severe depressive symptoms and a worse mental health outcome.
  units on a scale | 9.1 (5.6) | 9.1 (6.1) | 9.1 (5.8)
The Pain Catastrophizing Scale (PCS) [Mean (Standard Deviation); unit: units on a scale] — The Pain Catastrophizing Scale (PCS) is a 13-item self-report measure assessing exaggerated negative thoughts and feelings about pain. Each item is rated from 0 to 4, with the total score (0-52) calculated by summing all responses. Higher scores indicate greater pain catastrophizing and worse psychological outcomes related to pain.
  units on a scale | 39.8 (13.5) | 39.9 (14.0) | 39.8 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI) Total Score
Description: The Brief Pain Inventory (BPI) is a validated tool measuring pain severity and its impact on daily functioning. It includes 11 items assessing pain severity (worst, least, average, current) and pain interference with general activity, mood, walking, work, relations with others, sleep, and enjoyment of life. Each item is rated from 0 (no pain/no interference) to 10 (worst pain imaginable/complete interference). The Pain Severity Subscore (0-10) is the average of four severity items, the Functional Interference Subscore (0-10) is the average of seven interference items, and the Total Score (0-10) is the average of all 11 items. Higher scores indicate worse pain severity and greater pain interference.
Time Frame: Immediately postintervention and 3-month follow-up (postintervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills to Manage Pain (STOMP) | Comparison Group
Number analyzed (Participants) | 139 | 139
score on a scale
  Immediately postintervention | 4.74 (0.19) | 5.99 (0.19)
  3-month follow-up | 5.13 (0.19) | 5.74 (0.19)

2. Secondary Outcome: Brief Pain Inventory (BPI) Functional Interference Subscore
Description: as for outcome 1
Time Frame: Immediately postintervention and 3-month follow-up (postintervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills to Manage Pain (STOMP) | Comparison Group
Number analyzed (Participants) | 139 | 139
score on a scale
  Immediately postintervention | 4.41 (0.23) | 5.93 (0.23)
  3-month follow-up | 4.92 (0.24) | 5.57 (0.23)

3. Secondary Outcome: Brief Pain Inventory (BPI) Pain Severity Subscore
Description: as for outcome 1
Time Frame: Immediately postintervention and 3-month follow-up (postintervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills to Manage Pain (STOMP) | Comparison Group
Number analyzed (Participants) | 139 | 139
score on a scale
  Immediately postintervention | 5.13 (0.2) | 6.23 (0.19)
  3-month follow-up | 5.25 (0.2) | 6.11 (0.2)

4. Secondary Outcome: The Pain, Enjoyment and General Activity (PEG) Scale
Description: The Pain, Enjoyment and General Activity (PEG) scale measures pain severity and enjoyment of activities with scores ranging from 0 to 10. Higher scores indicate worse pain and greater interference with daily activities. The total score is the average of 3 items assessing pain intensity, enjoyment of life, and general activity.
Time Frame: Immediately postintervention and 3-month follow-up (postintervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills to Manage Pain (STOMP) | Comparison Group
Number analyzed (Participants) | 139 | 139
score on a scale
  Immediately postintervention | 5.61 (0.21) | 6.94 (0.2)
  3-month follow-up | 5.68 (0.21) | 6.78 (0.21)

5. Secondary Outcome: The Pain Self-Efficacy Questionnaire (PSEQ)
Description: The Pain Self-Efficacy Questionnaire (PSEQ) assesses an individual's confidence in their ability to perform daily activities despite pain. The total score is the sum of 10 items, each rated from 0 to 6, resulting in a range of 0 to 60. Higher scores indicate greater self-efficacy and a stronger belief in one's ability to manage daily tasks while experiencing pain.
Time Frame: Immediately postintervention and 3-month follow-up (postintervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills to Manage Pain (STOMP) | Comparison Group
Number analyzed (Participants) | 139 | 139
score on a scale
  Immediately postintervention | 40.53 (1.31) | 36.44 (1.28)
  3-month follow-up | 40.73 (1.33) | 35.91 (1.31)

6. Secondary Outcome: The Patient Health Questionnaire-8 (PHQ-8)
Description: The Patient Health Questionnaire-8 (PHQ-8) is an 8-item self-report measure assessing depressive symptoms over the past two weeks. Each item is rated from 0 to 3, with the total score (0-24) calculated by adding all responses, with higher scores indicating more severe depressive symptoms and a worse mental health outcome.
Time Frame: Immediately postintervention and 3-month follow-up (postintervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills to Manage Pain (STOMP) | Comparison Group
Number analyzed (Participants) | 139 | 139
score on a scale
  Immediately postintervention | 6.39 (0.48) | 8.66 (0.47)
  3-month follow-up | 7.25 (0.48) | 7.69 (0.48)

7. Secondary Outcome: The Pain Catastrophizing Scale (PCS)
Description: The Pain Catastrophizing Scale (PCS) is a 13-item self-report measure assessing exaggerated negative thoughts and feelings about pain. Each item is rated from 0 to 4, with the total score (0-52) calculated by summing all responses. Higher scores indicate greater pain catastrophizing and worse psychological outcomes related to pain.
Time Frame: Immediately postintervention and 3-month follow-up (postintervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills to Manage Pain (STOMP) | Comparison Group
Number analyzed (Participants) | 139 | 139
score on a scale
  Immediately postintervention | 34.35 (1.46) | 38.57 (1.44)
  3-month follow-up | 34.24 (1.48) | 35.99 (1.46)

ADVERSE EVENTS:
Time Frame: 2 years, 7 months
Description: Participants reported adverse events (AEs) during routine assessments and indicated if they were study-related. Study-related AEs were adjudicated by the site PI. All AEs were reported and reviewed in meetings. Events were classified by type (hospitalization, illness, injury) and grouped by severity: mild, moderate, severe, or very severe (see Adverse Event Term Additional Description). AEs were recorded based on participant descriptions rather than predefined Adverse Event Terms.
Arm/Group | Skills to Manage Pain (STOMP) | Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/139
Serious Adverse Events (participants affected / at risk) | 39/139 | 45/139
Other Adverse Events (participants affected / at risk) | 51/139 | 52/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Skills to Manage Pain (STOMP) (N=139) | Comparison Group (N=139)
Very Severe (General disorders) | 4 (4) | 7 (7) — Life-threatening, disabling, fatal event
Severe (General disorders) | 35 (35) | 38 (38) — Event required extensive medical attention; unable to carry out normal activities.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Skills to Manage Pain (STOMP) (N=139) | Comparison Group (N=139)
Moderate (General disorders) | 30 (30) | 34 (34) — Event resolved with treatment; normal activities conducted with some limitations.
Mild (General disorders) | 21 (21) | 18 (18) — Event required no or minimal treatment; able to carry out normal activities

LIMITATIONS AND CAVEATS:
Limitations include a specific population (people with HIV and chronic pain), limiting generalizability to other groups. Short follow-up (3 months) restricts insight into long-term effects. Women were slightly underrepresented, reducing applicability to chronic pain populations where women are more common. Participants were not blinded, possibly introducing bias, though staff and investigators remained blinded. Addressing these in future trials can improve applicability and robustness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03692611/Prot_SAP_001.pdf